CLINICAL TRIAL: NCT06094413
Title: The Effects of an 8-week Multicomponent Training Program on Quality of Life, Fear of Falling, &Amp; Physical Performance in Community-Dwelling Older Adults
Brief Title: Effects of Multicomponent Training in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-1091
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Sarcopenia
Keywords: Multicomponent Physical Activity; Older Adult; Quality of Life; Fear of Falling; Physical Performance
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Intervention Model Description: A mixed-methods study design was used to assess the effectiveness of a multicomponent training program on quality of life, fear of falling, and physical performance in older adults. The study included a pre-mid-post-test design with an intervention group who performed an 8-week multicomponent training program and a control group composed of patients who do not perform the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multicomponent Training Intervention (Experimental): Subjects in the intervention group attended two standardized group-based sixty-minute sessions per week in the outpatient medical center and were asked not to change their current physical activity regimen during the 8-week duration of the study.
  Interventions: Behavioral: Multicomponent Training Intervention
- Control Group (No Intervention): Subjects in the control group were asked to not change their current level of physical activity during the 8-week duration of the study.

INTERVENTIONS:
Behavioral: Multicomponent Training Intervention — The intervention was implemented and supervised by a well-trained, highly experienced professional with post-graduate education in the fields of exercise science and health promotion. Each session consisted of three phases: warm-up/initiation, conditioning, and cooldown. The intervention was composed of aerobic, resistance, balance, and flexibility exercises. At each session subjects werre informed of the program goals and the methods used to document exercise tolerance of the session's training loads. The quality of the intervention was measured by patient compliance, adherence, and feedback such as rates of perceived exertion (RPE) which were monitored during the session to measure immediate effect of the intervention. Progressions were guided by individual responsiveness and measured by RPE. Progressions were based on the training principles of specificity, adaptability, and overload.
  Arms: Multicomponent Training Intervention

SUMMARY:
The purpose of the study was to determine whether community-dwelling older adults would experience improved patient-reported outcomes and physical performance after completing an 8-week multicomponent exercise training program when compared to a control group who did not complete the intervention. As an additional aim, subjects who participated in the exercise intervention were asked about their experiences to identify factors that contributed to positive health behaviors in community-dwelling older adults.

DETAILED DESCRIPTION:
Sarcopenia is a geriatric syndrome which involves the progressive loss of muscle mass and physical performance in aging adults. The age-related decline inherent to sarcopenia has been associated with an increased risk of falls, disability, and mortality. Exercise is a non-pharmacological intervention that has been shown to prevent and manage age-related loss of muscle mass and strength, however there is limited research regarding its effect on patient-reported outcomes in older adults.

The purpose of this study is to examine the effects of an 8-week multicomponent training program on quality of life, fear of falling, and physical performance in community-dwelling older adults. A convenient sample of community-dwelling older adults aged 65 years and older from an outpatient medical center in Northeast Pennsylvania were recruited to participate. Eligible subjects volunteered to participate in the intervention, which consisted of two group-based sixty-minute standardized sessions per week supervised by an experienced professional in the outpatient medical center, or a control group composed of patients who did not perform the intervention. Outcomes testing was performed for both groups prior to, at the mid-point (4 weeks), and following the completion of the exercise intervention (8 weeks). Semi-structured, individual interviews with selected participants who completed the intervention were conducted by the researcher in the designated research environment to assess barriers, drivers, and the overall experience of the intervention.

The study evaluated the following research questions:

1. Will an 8-week multicomponent exercise intervention improve quality of life in community-dwelling older adults with probable sarcopenia?
2. Will an 8-week multicomponent exercise intervention improve fear of falling in community-dwelling older adults with probable sarcopenia?
3. Will an 8-week multicomponent exercise intervention improve physical performance in community-dwelling older adults with probable sarcopenia?
4. Will an 8-week multicomponent exercise intervention improve hand grip strength in community-dwelling older adults with probable sarcopenia?
5. What are the drivers and barriers of exercise adherence for community-dwelling older adults with probable sarcopenia who experienced an 8-week multicomponent exercise intervention?

A two-way ANOVA (group x time) was utilized for data analysis to determine between-group effects. Tukey post hoc testing was used to evaluate where differences occurred (pre-, mid-, post-). General ideas and emerging themes were inductively coded by the researcher and an independent content specialist utilizing the data from post-intervention interview transcripts.

The study was significant because it assessed whether the program was a feasible intervention that could be implemented by providers to aid in the management of age-related loss of muscle strength and physical performance for community-dwelling older adults. The findings of this study offered providers evidence-based practices that could be used for effective multicomponent exercise training prescription.

ELIGIBILITY:
Inclusion Criteria:

* age greater than or equal to 65 years
* able and willing to provide consent
* patient of Geisinger 65Forward Scranton clinic

Exclusion Criteria:

* Diagnosis of mild cognitive impairment, neurological disorders, uncontrolled metabolic disease, history of pacemaker or cardiovascular disease or high blood pressure not controlled with medication
* Previous history of musculoskeletal surgery or injury that could affect mobility
* An inability to perform an exercise program independently

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Short Physical Performance Battery (SPPB) composite score | Prior to the start of the intervention (Week 1), Mid-point of the intervention (Week 4), Following the completion of the Intervention (Week 8)
  The SPPB was utilized to measure physical performance in the present study. The SPPB is a valid and reliable tool for assessing lower extremity function and mobility in community-dwelling adults. The SPPB score measures lower extremity functional performance among older adults by assessing chair stand time, gait speed, and standing balance. SPPB scores range from zero (worst performance) to twelve (best performance) possible points.
Falls Efficacy Scale (FES) score | Prior to the start of the intervention (Week 1), Mid-point of the intervention (Week 4), Following the completion of the Intervention (Week 8)
  The FES is a tool that was developed to assess self-confidence while performing physical activity in conjunction with a fear of falling.The questionnaire addressed a patient's confidence in carrying out 10 daily tasks without falling. The FES score ranged from 10 (highest level of confidence) to 100 (lowest level of confidence) points. A score of greater than 80 indicates an increased risk of falling. A score of greater than 70 indicates a fear of falling.
Sarcopenia Quality of Life (SarQoL) score | Prior to the start of the intervention (Week 1), Mid-point of the intervention (Week 4), Following the completion of the Intervention (Week 8)
  The SarQoL is a patient-reported outcome measurement (PROM) designed to assess quality of life in individuals aged 65 years and older who have been diagnosed with sarcopenia. It is a self-administered questionnaire including 22 questions, rated on a 4-point Likert scale. It assessed perceived domains such as physical and mental health, fears, and functionality in daily life. Each domain was scored from 0-100 and an Overall Score was calculated. The total scoring ranged from 0(worst imaginable health) to 100 (best imaginable health).

SECONDARY OUTCOMES:
Hand Grip Strength score | Pre-intervention during the screening process, Mid-point of the intervention (Week 4), Following the completion of the Intervention (Week 8)
  A hand dynamometer was used to assess hand grip strength in both upper extremities. The instrument score was calculated in kg (0-90) with a lower score indicating lower hand grip strength and a higher score indicating higher hand grip strength.

OTHER OUTCOMES:
Qualitative Data from semi-structured interviews | Following completion of the intervention (Week 8)
  Post-intervention interviews were completed after completion of the 8-week intervention by willing subjects to identify drivers, barriers, and satisfaction levels for participants. Interviews were 15 minutes in length, held in the same area as the intervention, recorded through Zoom communication platform, and then transcribed for qualitative analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Goodrich, DO, Principal Investigator — Geisinger Clinic; Shala Davis, PhD, Study Chair — East Stroudsburg University
Locations (1):
- Geisinger 65Forward, Scranton, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tinetti ME, Richman D, Powell L. Falls efficacy as a measure of fear of falling. J Gerontol. 1990 Nov;45(6):P239-43. doi: 10.1093/geronj/45.6.p239. PMID 2229948
- [Background] American Psychological Association. (2023). Mild cognitive impairment. In APA dictionary of psychology. https://dictionary.apa.org/mild-cognitive-impairment
- [Background] Beaudart C, Biver E, Reginster JY, Rizzoli R, Rolland Y, Bautmans I, Petermans J, Gillain S, Buckinx F, Dardenne N, Bruyere O. Validation of the SarQoL(R), a specific health-related quality of life questionnaire for Sarcopenia. J Cachexia Sarcopenia Muscle. 2017 Apr;8(2):238-244. doi: 10.1002/jcsm.12149. Epub 2016 Oct 22. PMID 27897430
- [Background] Bohannon RW. Minimal clinically important difference for grip strength: a systematic review. J Phys Ther Sci. 2019 Jan;31(1):75-78. doi: 10.1589/jpts.31.75. Epub 2019 Jan 10. PMID 30774209
- [Background] Chen LK, Woo J, Assantachai P, Auyeung TW, Chou MY, Iijima K, Jang HC, Kang L, Kim M, Kim S, Kojima T, Kuzuya M, Lee JSW, Lee SY, Lee WJ, Lee Y, Liang CK, Lim JY, Lim WS, Peng LN, Sugimoto K, Tanaka T, Won CW, Yamada M, Zhang T, Akishita M, Arai H. Asian Working Group for Sarcopenia: 2019 Consensus Update on Sarcopenia Diagnosis and Treatment. J Am Med Dir Assoc. 2020 Mar;21(3):300-307.e2. doi: 10.1016/j.jamda.2019.12.012. Epub 2020 Feb 4. PMID 32033882
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Background] de Fatima Ribeiro Silva C, Ohara DG, Matos AP, Pinto ACPN, Pegorari MS. Short Physical Performance Battery as a Measure of Physical Performance and Mortality Predictor in Older Adults: A Comprehensive Literature Review. Int J Environ Res Public Health. 2021 Oct 10;18(20):10612. doi: 10.3390/ijerph182010612. PMID 34682359
- [Background] Delbaere K, Close JC, Mikolaizak AS, Sachdev PS, Brodaty H, Lord SR. The Falls Efficacy Scale International (FES-I). A comprehensive longitudinal validation study. Age Ageing. 2010 Mar;39(2):210-6. doi: 10.1093/ageing/afp225. Epub 2010 Jan 8. PMID 20061508
- [Background] de Mello RGB, Dalla Corte RR, Gioscia J, Moriguchi EH. Effects of Physical Exercise Programs on Sarcopenia Management, Dynapenia, and Physical Performance in the Elderly: A Systematic Review of Randomized Clinical Trials. J Aging Res. 2019 Nov 20;2019:1959486. doi: 10.1155/2019/1959486. eCollection 2019. PMID 31827927
- [Background] Dismore L, Hurst C, Sayer AA, Stevenson E, Aspray T, Granic A. Study of the Older Adults' Motivators and Barriers Engaging in a Nutrition and Resistance Exercise Intervention for Sarcopenia: An Embedded Qualitative Project in the MIlkMAN Pilot Study. Gerontol Geriatr Med. 2020 May 19;6:2333721420920398. doi: 10.1177/2333721420920398. eCollection 2020 Jan-Dec. PMID 32490038
- [Background] Fielding RA, Rejeski WJ, Blair S, Church T, Espeland MA, Gill TM, Guralnik JM, Hsu FC, Katula J, King AC, Kritchevsky SB, McDermott MM, Miller ME, Nayfield S, Newman AB, Williamson JD, Bonds D, Romashkan S, Hadley E, Pahor M; LIFE Research Group. The Lifestyle Interventions and Independence for Elders Study: design and methods. J Gerontol A Biol Sci Med Sci. 2011 Nov;66(11):1226-37. doi: 10.1093/gerona/glr123. Epub 2011 Aug 8. PMID 21825283
- [Background] Geerinck A, Alekna V, Beaudart C, Bautmans I, Cooper C, De Souza Orlandi F, Konstantynowicz J, Montero-Errasquin B, Topinkova E, Tsekoura M, Reginster JY, Bruyere O. Standard error of measurement and smallest detectable change of the Sarcopenia Quality of Life (SarQoL) questionnaire: An analysis of subjects from 9 validation studies. PLoS One. 2019 Apr 29;14(4):e0216065. doi: 10.1371/journal.pone.0216065. eCollection 2019. PMID 31034498
- [Background] Geriatrics. American Physical Therapy Association (APTA). (2021). Outcome measure toolkit for geriatric fall/balance assessment. https://www.aptageriatrics.org/special-interest-groups/balance-falls/Outcome-Measure-Toolkit/Outcome%20Measures%20Toolkit%202020.pdf
- [Background] Hecksteden A, Faude O, Meyer T, Donath L. How to Construct, Conduct and Analyze an Exercise Training Study? Front Physiol. 2018 Jul 26;9:1007. doi: 10.3389/fphys.2018.01007. eCollection 2018. PMID 30140237
- [Background] Jenkins NDM, Cramer JT. Reliability and Minimum Detectable Change for Common Clinical Physical Function Tests in Sarcopenic Men and Women. J Am Geriatr Soc. 2017 Apr;65(4):839-846. doi: 10.1111/jgs.14769. Epub 2017 Mar 15. PMID 28295148
- [Background] Kaushal N, Langlois F, Desjardins-Crepeau L, Hagger MS, Bherer L. Investigating dose-response effects of multimodal exercise programs on health-related quality of life in older adults. Clin Interv Aging. 2019 Jan 24;14:209-217. doi: 10.2147/CIA.S187534. eCollection 2019. PMID 30774322
- [Background] Kumar P, Umakanth S, Girish N. A review of the components of exercise prescription for sarcopenic older adults. Eur Geriatr Med. 2022 Dec;13(6):1245-1280. doi: 10.1007/s41999-022-00693-7. Epub 2022 Sep 2. PMID 36050581
- [Background] Liguori, G. (2021). ACSM's Guidelines for Exercise Testing and Prescription, 11th Edition.
- [Background] Makizako H, Nakai Y, Tomioka K, Taniguchi Y, Sato N, Wada A, Kiyama R, Tsutsumimoto K, Ohishi M, Kiuchi Y, Kubozono T, Takenaka T. Effects of a Multicomponent Exercise Program in Physical Function and Muscle Mass in Sarcopenic/Pre-Sarcopenic Adults. J Clin Med. 2020 May 8;9(5):1386. doi: 10.3390/jcm9051386. PMID 32397192
- [Background] Malmstrom TK, Miller DK, Simonsick EM, Ferrucci L, Morley JE. SARC-F: a symptom score to predict persons with sarcopenia at risk for poor functional outcomes. J Cachexia Sarcopenia Muscle. 2016 Mar;7(1):28-36. doi: 10.1002/jcsm.12048. Epub 2015 Jul 7. PMID 27066316
- [Background] Phu S, Kirk B, Bani Hassan E, Vogrin S, Zanker J, Bernardo S, Duque G. The diagnostic value of the Short Physical Performance Battery for sarcopenia. BMC Geriatr. 2020 Jul 13;20(1):242. doi: 10.1186/s12877-020-01642-4. PMID 32660438
- [Background] Rizzoli R, Reginster JY, Arnal JF, Bautmans I, Beaudart C, Bischoff-Ferrari H, Biver E, Boonen S, Brandi ML, Chines A, Cooper C, Epstein S, Fielding RA, Goodpaster B, Kanis JA, Kaufman JM, Laslop A, Malafarina V, Manas LR, Mitlak BH, Oreffo RO, Petermans J, Reid K, Rolland Y, Sayer AA, Tsouderos Y, Visser M, Bruyere O. Quality of life in sarcopenia and frailty. Calcif Tissue Int. 2013 Aug;93(2):101-20. doi: 10.1007/s00223-013-9758-y. Epub 2013 Jul 5. PMID 23828275
- [Background] Safonova, Y. A. (2020). Sarcopenia risk factor for falls and fractures. The Clinician, 13(3-4), 22-28. https://doi.org/10.17650/1818-8338-2019-13-3-4-22-28
- [Background] Slade SC, Dionne CE, Underwood M, Buchbinder R. Consensus on Exercise Reporting Template (CERT): Explanation and Elaboration Statement. Br J Sports Med. 2016 Dec;50(23):1428-1437. doi: 10.1136/bjsports-2016-096651. Epub 2016 Oct 5. PMID 27707738
- [Background] Tsekoura M, Billis E, Tsepis E, Dimitriadis Z, Matzaroglou C, Tyllianakis M, Panagiotopoulos E, Gliatis J. The Effects of Group and Home-Based Exercise Programs in Elderly with Sarcopenia: A Randomized Controlled Trial. J Clin Med. 2018 Nov 26;7(12):480. doi: 10.3390/jcm7120480. PMID 30486262
- [Background] U.S. Department of Health & Human Services. (2018). Physical Activity Guidelines for Americans, 2nd edition. https://health.gov/sites/default/files/2019-09/Physical_Activity_Guidelines_2nd_edition.pdf
- [Background] Witham MD. Bridging the gap between the laboratory and the clinic for patients with sarcopenia. Biogerontology. 2019 Apr;20(2):241-248. doi: 10.1007/s10522-018-09793-z. Epub 2018 Dec 27. PMID 30591980
- [Background] Xia L, Zhao R, Wan Q, Wu Y, Zhou Y, Wang Y, Cui Y, Shen X, Wu X. Sarcopenia and adverse health-related outcomes: An umbrella review of meta-analyses of observational studies. Cancer Med. 2020 Nov;9(21):7964-7978. doi: 10.1002/cam4.3428. Epub 2020 Sep 13. PMID 32924316